CLINICAL TRIAL: NCT02966769
Title: Multicentric Retrospective Observation Study: Neoadjuvant Treatment and Surgery Versus Definitive Chemoradiation in the Non-Small Cell Lung Cancer (NSCLC) IIIA-N2
Brief Title: N2 Lung Cancer Project: Neoadjuvant Treatment Followed Surgery Versus Chemoradiation
Status: Completed | Type: Observational
Sponsor: Grupo de Investigación Clínica en Oncología Radioterapia (Other)
Responsible Party: Principal Investigator, Felipe Couñago, Doctor, Grupo de Investigación Clínica en Oncología Radioterapia
Other Study IDs: GICOR -SEOR 5-16
Record Dates: First submitted 2016-11-11; First posted 2016-11-17 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Non-small-Cell Lung Carcinoma; Surgery; Stage IIIA-N2; Chemoradiation; Survival
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chemoradiation Group: Analyze overall survival in the group of patients treatment by Concurrent Radiotherapy (>/= 60 Gy) plus Platinum-based Chemotherapy
  Interventions: Other: Overall survival
- Neoadjuvant treatment plus Surgery Group: Analyze overall survival in the group of patients treatment by Neoadjuvant Platinum-based Chemotherapy or Chemoradiation (Platinum-based plus >/= 45Gy) followed by Surgery
  Interventions: Other: Overall survival

INTERVENTIONS:
Other: Overall survival — Compare overall survival between both groups.

SUMMARY:
The objective of this multicenter retrospective study is to compare overall survival in patients with stage IIIA-N2 NSCLC treated with neoadjuvant treatment and surgery versus definitive chemoradiation.

Secondary objectives are to analyze disease-free survival, median survival, locoregional and distant relapses as well as mortality and toxicity related to treatment.

DETAILED DESCRIPTION:
Based on data published by the Intergroup 0139 trial, induction therapy followed by surgery in patients with stage IIIA-N2 NSCLC can increase overall survival compared to exclusive radical chemoradiation treatment.

The major handicap of all studies addressing the role of surgery in IIIA-N2 NSCLC is the difficulty of recruiting patients. Therefore, multicenter studies are necessary to confirm the hypothesis generated by the INT 0139.

ELIGIBILITY:
Inclusion Criteria:

* Stage IIIA (N2) disease
* Potentially resectable disease
* Stage Lung Cancer with CT scan or PET-CT.
* N2 involvement: it is not necessary pathological proof.
* No progression after induction treatment.

Exclusion Criteria:

* T4 or N3 stage.
* Bulky disease or not resectable.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with stage IIIA-N2 NSCLC potentially resectable at diagnosis.
Sampling Method: Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2016-06; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5 years

SECONDARY OUTCOMES:
Disease-free survival | 5 years
Patterns of Relapse | 5 years
Mortality | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Couñago, MD PhD, Principal Investigator — Grupo de Investigación Clínica en Oncología Radioterapia; Sara Montemuiño, MDPhd, Principal Investigator — Grupo de Investigación Clínica en Oncología Radioterapia
Locations (1):
- Hospital Universitario Quiron Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No